CLINICAL TRIAL: NCT02125097
Title: Multi-center Non-randomized Clinical Investigation of the Reverse Medical Barrel™ Vascular Reconstruction Device (VRD) for Adjunctive Treatment to Embolic Coils for Wide Neck Intracranial Bifurcation and Branch Aneurysms
Brief Title: The Reverse Barrel™ VRD Intracranial Aneurysm Trial
Acronym: Barrel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Barrel OUS VRD-001
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Intracranial Aneurysms
Keywords: Intracranial Aneurysm Treatment; Endovascular Therapy
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intracranial Aneurysm Treatment (Experimental): Barrel™ Vascular Reconstruction Device (VRD) is Intended for use with embolic coils for the treatment of wide-neck bifurcating or branch intracranial aneurysms arising from a parent vessel with a diameter of ≥ 2.0 mm and ≤ 4 mm, measured by 2D Digital Subtraction Angiography (DSA). Wide-neck is defined as having a neck width ≥ 4 mm or a dome-to-neck ratio < 2.
  Interventions: Device: Barrel™ Vascular Reconstruction Device (VRD)

INTERVENTIONS:
Device: Barrel™ Vascular Reconstruction Device (VRD) — Intended for use with embolic coils for the treatment of wide-neck bifurcating or branch intracranial aneurysms arising from a parent vessel with a diameter of ≥ 2.0 mm and ≤ 4 mm, measured by 2D Digital Subtraction Angiography (DSA). Wide-neck is defined as having a neck width ≥ 4 mm or a dome-to-neck ratio < 2.

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and effectiveness of the Barrel™ VRD when used to facilitate endovascular coiling of wide-neck bifurcating or branch intracranial aneurysms with any approved embolic coils.

ELIGIBILITY:
Summary Inclusion Criteria:

1. Male or female ≥18 years old.
2. A wide neck, intracranial, bifurcating or branch aneurysm with a neck ≥4 mm or a dome-to-neck ratio <2, including non-de novo aneurysms where no stent was utilized.
3. Subject's aneurysm arises from a parent vessel with a diameter ≥ 2.0 mm and ≤ 4mm, measured by 2D Digital Subtraction Angiography (DSA).
4. Subject responds to anti-coagulation and anti-platelet therapy according to the test used in each study center.
5. Subject is eligible to undergo a procedure with the use of contrast media.
6. Subject is willing to comply with protocol requirements and return to the treatment center for all required clinical evaluations and follow-up.
7. Subject has given written informed consent.
8. Life expectancy > 12 months.

   -

Summary Exclusion Criteria:

1. Subject presents with ruptured aneurysm, unless rupture occurred 30 days or more prior to screening.
2. Subject is currently undergoing radiation therapy.
3. Subject has known allergies to nickel-titanium metal.
4. Subject has known allergies to aspirin, heparin, ticlopidine, or clopidogrel.
5. Subject has a life-threatening allergy to contrast media (unless treatment for allergy can be tolerated).
6. Subject has a known cardiac disorder, likely to be associated with cardio-embolic symptoms such as atrial fibrillation (AFIB).
7. Subject has any condition, which in the opinion of the treating physician, would place the subject at a high risk of embolic stroke.
8. Subject is currently participating in another clinical research study.
9. Subject has had a previous intracranial stenting procedure associated with the target aneurysm.
10. Subject is unable to complete the required follow-up.
11. Subject is pregnant or breastfeeding.(Females of childbearing potential must have a pregnancy test and provide written proof that they are not pregnant prior to inclusion.)
12. Subject has participated in a drug study within the last 30 days.
13. Subject who cannot or is unwilling to take ASA/Clopidogrel for a minimum of at least 3 months following the procedure.
14. Extradural aneurysms.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2015-12-12 (Actual); Study Completion 2015-12-12 (Actual)

PRIMARY OUTCOMES:
Successful aneurysm occlusion with the Barrel™ VRD, as measured by angiography with an aneurysm Raymond Grade Scale of 1 or 2 at 12 months post procedure | 12 months
  Effectiveness measures are successful aneurysm treatment with the Barrel™ VRD, as measured by angiography with an aneurysm Raymond Grade Scale of 1 or 2 at 12 months post procedure in the absence of retreatment, parent artery stenosis (> 50%), or target aneurysm rupture.
  Safety measures are the absence of neurological death or major stroke at 12 months post treatment.

SECONDARY OUTCOMES:
Successful delivery of the device measured by technical success. | At implant up to 30 days
  Technical success is defined as access to the lesion, successful deployment of the Barrel™ VRD and correct positioning of the device over the aneurysm.

OTHER OUTCOMES:
Functional outcome | At 12 months
  Functional outcome as defined by modified Rankin Scale (mRS) at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Piotin, M.D., Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild, Paris, France
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Gory B, Blanc R, Turjman F, Berge J, Piotin M. The Barrel vascular reconstruction device for endovascular coiling of wide-necked intracranial aneurysms: a multicenter, prospective, post-marketing study. J Neurointerv Surg. 2018 Oct;10(10):969-974. doi: 10.1136/neurintsurg-2017-013602. Epub 2018 Feb 2. PMID 29437935